CLINICAL TRIAL: NCT04441411
Title: Non Fusion Surgery in Adolescent Idiopathic Scoliosis Patients Using the Nemost-AIS System
Brief Title: Non Fusion Surgery in Adolescent Idiopathic Scoliosis Patients
Acronym: NEMOST-AIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, BJ van Royen, clinical professor, principal investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL67124.018.19; NL8659 (Other: NTR)
Record Dates: First submitted 2020-06-11; First posted 2020-06-22 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: scoliosis; nonfusion; surgery; fusionless; idiopathic; adolescent
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NEMOST-AIS (Other): This study is designed as a cohort study.
  Interventions: Device: NEMOST system

INTERVENTIONS:
Device: NEMOST system — Minimal invasive double rod posterior Non-Fusion Scoliosis Surgery

SUMMARY:
The primary objective of the study is to monitor the effectiveness of a minimal invasive non-fusion double rod bipolar posterior spinal implant (Nemost growing domino) to correct the scoliotic curve in growing patients suffering from progressive adolescent idiopathic scoliosis (AIS) who have failed conservative treatment.

DETAILED DESCRIPTION:
Scoliosis is a complex three-dimensional deformity of the spine, which occurs primarily in growing children and adolescents. In adolescent idiopathic scoliosis (AIS), the cause is unknown. Children with severe and progressive scoliosis, if left untreated, are at risk of rapid and severe spinal deformity progression, which can result in a decrease of pulmonary function, poor cosmetic result and poor quality of life.

Treatment options in AIS depend on curve severity and remaining growth potential, and include intensive brace treatment for smaller curvatures whereas surgical correction and spinal fusion is advocated for more severe curves. Growing rods are used for severe early infantile deformities or early onset scoliosis (EOS).

Bracing, by using a rigid plastic orthosis, is currently the primary therapy to prevent curve progression in mild curves up to 45 degrees and skeletal immature patients. Most braces are recommended to be worn for 18-23 hours per day during several years (until skeletal maturity has been reached). This may cause a high level of physical discomfort and emotional and psychological stress in these patients, and failure of brace treatment therefore is common.

Surgical therapy for AIS is recommended in severe progressive curvatures. Surgical treatment includes correction of the spinal curvature by using multisegmental screw fixation and posterior spinal fusion of the thoracolumbar spine. Complete posterior spinal fusion, however, lacks the possibilities for future adaptation of natural changes in spinal balance and posture.

Currently, growing rods systems are used as a posterior spinal implant to allow growth of the spine and thorax and limit progression of the scoliosis in young patients with early onset scoliosis. Growing rods systems are distractible spinal implants, with bipolar anchorage fixations to the upper and lower part of the spine, using posterior spinal instrumentation such as hooks and pedicle screws.

The Nemost growing system, developed by the EUROS Compagny, is a CE-marked commercial available medical device for the treatment of early onset neuromuscular or early onset idiopathic scoliosis. It is a non-fusion, growth enabling system with bipolar fixation intended to be used with a posterior spinal instrumentation.

It is hypothesized that the use of a minimal invasive non-fusion bipolar posterior spinal implant (Nemost growing domino) can both correct and brace the spine internally and adapt balans and or distraction as the idiopathic scoliosis patient grows.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent idiopathic scoliosis ;
* Primary Cobb angle greater than 30°;
* Failed non-operative treatment defined as progression of the curve greater than 5° per year at any time;
* Skeletally immature (Risser grade* ≤2 and Skeletal age of hand and wrist X-rays ≤14y);
* In girl, either pre-menarchal or post-menarchal by no more than 1 year;
* Age over 10 years;
* Non rigid curve;
* All Lenke type;
* No previous spine surgery.

Exclusion Criteria:

* Non-idiopathic scoliosis: musculoskeletal or neurologic conditions responsible for cause of the spine curvature (i.e. neuromuscular, congenital or syndromic scoliosis);
* History of previous spine surgery;
* Risser sign >2;
* Disease or deformity likely to affect the stability of the device (i.e. inadequate anatomy of pedicles, trauma or tumor in fixation region, severe osteoporosis, bone destruction or poor bone quality);
* Non-reductible scoliosis;
* Known allergy or intolerance to one of the device material;
* Acute or chronic infections, local or systemic;
* Absence or insufficience of covering tissues;
* Pathological obesity.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2020-06-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Coronal balance (Correction of the primary curvature on radiograph | 2 years
  Cobb angle (degrees)
T1-S1 length on radiograph | 2 years
  length (cm)
instrument segment length on radiograph | 2 years
  length (cm)
(Serious) Adverse Event | 2 years
  complications
Sagittal balance (thoracic kyphosis, lumbar lordosis, proximal and distal junctional angle) | 2 years
  Cobb angle (degrees)
Pelvic parameters (pelvic obliquity, sacral slope, pelvic incidence, pelvic tilt) | 2 years
  degrees

SECONDARY OUTCOMES:
Vertebral rotation | 2 years
  scoliometer assesment
Patient Reported Outcome (PRO | 2 years
  Scoliosis Research Society's-22 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: BJ Van Royen, MD, PhD, Principal Investigator — AmsterdamUMC
Locations (1):
- AmsterdamUMC, location AMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Post AM, Berends HI, van Royen BJ. Minimally Invasive Posterior Spinal Nonfusion Surgery in Patients With Adolescent Idiopathic Scoliosis Using a Bipolar One-Way Self-Expanding Rod System: Protocol for a Single-Center Clinical Cohort Study. JMIR Res Protoc. 2023 Dec 25;12:e47222. doi: 10.2196/47222. PMID 38145474